CLINICAL TRIAL: NCT02453906
Title: Cerebral Response of Healthy Subjects to a Somatosensory Stimulation With XNKQ Acupuncture Compared to Control Interventions Measured With EEG and fMRI
Brief Title: XNKQ Acupuncture Compared to Control Interventions Measured With EEG and fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia M. Witt (Other)
Responsible Party: Sponsor-Investigator, Claudia M. Witt, Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: XNKQ-15
Record Dates: First submitted 2015-04-29; First posted 2015-05-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy subjects (Experimental): they receive XNKQ acupuncture, as well as control 1, control 2, and control 3 in a randomized order.
  Interventions: Other: XNKQ; Other: Control 1; Other: Control 2; Other: Control 3

INTERVENTIONS:
Other: XNKQ — stimulation at 5 acupuncture points according to XNKQ acupuncture
Other: Control 1 — no stimulation at 5 acupuncture points according to XNKQ acupuncture
Other: Control 2 — stimulation at 5 control points
Other: Control 3 — no stimulation at 5 control points

SUMMARY:
The investigators will use EEG, structural MRI, and resting-state functional connectivity MRI to assess neuronal responses in 28 healthy subjects to different somatosensory stimulations.

DETAILED DESCRIPTION:
To develop a better understanding of the cerebral response to a complex somatosensory intervention with XNKQ acupuncture and to build a foundation for future studies with stroke patients our study aims to evaluate changes of brain activity and brain structure in healthy subjects after XNKQ acupuncture in comparison to three control interventions. We will use EEG, structural MRI, and resting-state functional connectivity MRI to assess neuronal responses in 28 healthy subjects to a) strong manual needle-stimulation of the acupuncture points DU26, PC6 and SP6 (XNKQ acupuncture), b) insertion of needles on the acupuncture points DU26, PC6 and SP6 without stimulation (control 1), c) strong manual needle stimulation of three non-acupuncture points (control 2), and d) insertion of needles on three non-acupuncture points without stimulation (control 3). With this, our study aims to create results which inform future studies in patients and might be helpful for the rehabilitation of deficits after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (18 to 40 years of age) health status confirmed by a comprehensive neurological examination
* Right-handed (evaluated by "the Edinburgh inventory")
* Informed consent
* No acupuncture treatment in the last 12 months
* No medical knowledge about acupuncture

Exclusion Criteria:

* History of neurological and/or psychiatric diseases
* History of brain injury
* Cognitive handicap and severe speech disorder
* alcohol or drug abuse
* History of neurosurgical intervention
* Chronic disease (e.g., asthma, diabetes mellitus etc.) with regular use of medications
* Usage of acute medication
* Pregnancy (tested by urine pregnancy test before the measurement) or planned pregnancy
* Any contraindication for acupuncture (e.g., anti-coagulation therapy)
* Any exclusion criteria for MRI scanning (metal implants (e.g. pacemaker), claustrophobia, etc.)
* Participation in another interventional trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in brain background rhythms (mu-alpha and beta activity) [assessed using EEG and MRI] after one intervention (baseline vs. post stimulation) in comparison between the four different interventions. | 60 minutes
Changes in resting state functional connectivity [assessed using EEG and MRI] after one intervention (baseline vs. post-stimulation) in comparison between the four different interventions | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M. Witt, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Nierhaus T, Chang Y, Liu B, Shi X, Yi M, Witt CM, Pach D. Somatosensory Stimulation With XNKQ Acupuncture Modulates Functional Connectivity of Motor Areas. Front Neurosci. 2019 Mar 11;13:147. doi: 10.3389/fnins.2019.00147. eCollection 2019. PMID 30914909